CLINICAL TRIAL: NCT06967896
Title: A Randomized Controlled Trial Comparing Different Models of Tracheal Tube for Thyroid Surgery in Women
Brief Title: Different Models of Tracheal Catheters Are Used for Female Thyroid Glands
Status: Recruiting | Type: Observational
Sponsor: Anqing Municipal Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Sun LingLU
Record Dates: First submitted 2025-04-19; First posted 2025-05-13 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2024-10

CONDITIONS: Sore Throat; Tracheal Tubes With an Inner Diameter of 6.0mm; Tracheal Tubes With an Inner Diameter of 6.5mm; Tracheal Tubes With an Inner Diameter of 7.0mm
Keywords: thyroid surgery; sore throat; Tracheal tube
MeSH Terms: conditions — Pharyngitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- 6.0#: Insert the tracheal tube of model 6.0#
- 6.5#: Insert the tracheal tube of model 6.5#
- 7.0#: Insert the tracheal tube of model 7.0#

SUMMARY:
Objective:Compare whether the use of tracheal catheters of models 6.0 and 6.5 causes less sore throat in women after thyroid surgery compared with the traditional use of model 7.0 tracheal catheters.Methods: Investigators enrolled 180 female patients with American Society of Anesthesiologists (ASA) physical status I and III, aged 18-65 years, and scheduled for elective undergoing thyroid surgery with general anesthesia. The participants were randomly assigned into three groups(n=60 each group):Group A: Tracheal catheter group with an inner diameter of 6.0mm, Group B: Tracheal catheter group with an inner diameter of 6.5mm, Group C: Tracheal catheter group with an inner diameter of 7.0mm.The incidence and severity of postoperative sore throat were recorded in three groups at 1 h, 6 h, 24 h and 48 h after operation.

ELIGIBILITY:
Inclusion Criteria:

* Female;
* Thyroid surgery should be performed under general anesthesia (GA) at an appropriate time;
* ASA grade I-III;
* Aged 18-65 years;
* BMI less than 35Kg/m2
* In line with ethics, patients voluntarily accept this experiment and sign informed consent.

Exclusion Criteria:

* Reflux esophagitis, preoperative sore throat, chronic pharyngitis, preoperative hoarseness, use of anticoagulants or corticosteroids, high risk of reflux or aspiration, dysphagia, previous oral or pharyngeal surgical intervention, bleeding disorder, severe heart, lung, liver and kidney dysfunction
* Upper respiratory tract infection occurred within 2 weeks before surgery
* Unable to insert ET (no more than two intubations)
* Patients with hoarseness or sore throat before surgery
* Language communication, hearing impairment or brain dysfunction such as stroke, unable to communicate

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Healthy female thyroid surgery patients, ages 18-65 years, did not have serious systemic disease
Sampling Method: Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2024-10-09 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
The incidence of postoperative sore throat | at 1 hour, 6 hour, 24 hour and 48 hour after operation
  The incidence of postoperative sore throat

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anqing Hospital Anesthesiology, Anqing, Anhui, China

IPD SHARING:
Plan to Share IPD: No